CLINICAL TRIAL: NCT00589498
Title: Fat Gain and Cardiovascular Disease Mechanisms
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Virend Somers, Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 652-03; NIH HL-073211
Record Dates: First submitted 2008-01-07; First posted 2008-01-09 (Estimated); Last update posted 2013-11-04 (Estimated); Status verified 2013-11

CONDITIONS: Hypertension; Sleep Apnea Syndromes; Obesity
MeSH Terms: conditions — Hypertension; Sleep Apnea Syndromes; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Subjects who are randomized to overfeed will visit with the General Clinical Research Center dieticians as often as necessary to gain 2 kg of fat (about 4 kg overall) over a period of 8 weeks.
  Interventions: Dietary Supplement: 1000 extra calories
- 2 (No Intervention): Subjects who are randomized to non-overfeeding will continue with their normal diet and activity levels for a period of 8 weeks.

INTERVENTIONS:
Dietary Supplement: 1000 extra calories — Each subject received 1000 kcal/d in addition to weight maintenance requirements. The diet composition throughout the study was 40% carbohydrate, 40% fat, and 20% protein.
  Arms: 1

SUMMARY:
Understanding the mechanisms of obesity-induced hypertension is important both for prevention and therapy. Studies of patients with established obesity have provided valuable information on pathophysiologic links between obesity and both blood pressure and cardiovascular risk. However, these studies are necessarily limited by the heterogeneity of obesity-associated disease so that the relative contribution of obesity or hypertension or other co-existing diseases to specific regulatory abnormalities is often not clear. Clarification of whether any abnormalities associated with increased cardiovascular risk were present before or after the development of obesity has also been problematic.

We therefore propose a series of novel studies directed at establishing the effects of increased body fat in otherwise healthy individuals. We will determine the distribution patterns of increased body fat and how both increased body fat and fat distribution relate to changes in blood pressure, and in neural, endothelial and inflammatory mechanisms which have been implicated in the development and progression of cardiac and vascular disease.

We will study non-obese subjects with and without a family history of hypertension. These subjects will undergo an eight-week program of overfeeding with the objective of inducing a 4 kg fat gain. We will determine the nature of fat distribution in these individuals after the fat gain program and subsequently after an eight-week period of weight loss and restoration of normal body weight. Measurements will be compared to those obtained in a matched control group with and without a family history of hypertension, who will continue their normal diets. We will test the following hypotheses:

* Individuals with a family history of hypertension will gain more visceral fat and upper body subcutaneous fat and will have greater blood pressure increases with overfeeding- compared with those without such a family history.
* For all overfed subjects, increases in blood pressure and insulin resistance with fat gain will be most marked in those individuals with a predominantly upper body and visceral fat accumulation.
* Upper body and visceral fat gain will also be associated with greater impairment in cardiovascular function, higher nocturnal blood pressures and an increased likelihood of sleep disordered breathing.

ELIGIBILITY:
Inclusion Criteria:

* We will enroll up to 180 subject in order to fulfill screening requirements and have complete studies in 120 total (60 with and 60 without family history hypertension).
* Gender: Male and female.
* Ages: 18 to 40 (inclusive).

Exclusion Criteria:

* Body-mass index > 33 kg/m2
* Tobacco smoking or chewing
* Shift worker
* Any diseases
* Any prescription medications (except, oral contraceptives are permitted)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2005-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Individuals with a family history of hypertension will gain more visceral fat and upper body subcutaneous fat and will have greater blood pressure increases with overfeeding- compared with those without such a family history. | conclude the 180 patients recruited

SECONDARY OUTCOMES:
* For all overfed subjects, increases in blood pressure and insulin resistance with fat gain will be most marked in those individuals with a predominantly upper body and visceral fat accumulation. | after recruiting at least 70 patients
Upper body and visceral fat gain will also be associated with greater impairment in cardiovascular function, higher nocturnal blood pressures and an increased likelihood of sleep disordered breathing | Recruit at least 70 subjects
Increased weight gain, particularly in the upper body and visceral regions, will be accompanied by enhanced production of inflammatory mediators linked to cardiovascular risk, including adhesion molecules and C-reactive protein. | Recruit at least 70 patients
These changes will resolve with subsequent loss of weight at the end of the overfeeding program and restoration of normal body fat and fat distribution. | Recruit at least 70 patients

CONTACTS AND LOCATIONS:
Overall Officials: Virend K Somers, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Romero-Corral A, Sert-Kuniyoshi FH, Sierra-Johnson J, Orban M, Gami A, Davison D, Singh P, Pusalavidyasagar S, Huyber C, Votruba S, Lopez-Jimenez F, Jensen MD, Somers VK. Modest visceral fat gain causes endothelial dysfunction in healthy humans. J Am Coll Cardiol. 2010 Aug 17;56(8):662-6. doi: 10.1016/j.jacc.2010.03.063. PMID 20705223